CLINICAL TRIAL: NCT07329179
Title: Crestal Sinus Lifting Using Densah Burs Versus Lateral Window Technique at Residual Alveolar Ridge Height 3-5 mm With Simultaneous Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A02061222
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sinus Pneumatization
Keywords: Densah burs, CBCT, Sinus lifting, Implant

STUDY DESIGN:
Intervention Model Description: The patients were divided randomly into two equal groups; each included 7 implants:
  - For group I: Sinus membrane elevation procedure using densah burs with crestal approach followed by bone grafting and simultaneous implant placement were done in this group.
  - For group II: Sinus membrane elevation procedure using lateral window technique followed by bone grafting and simultaneous implant placement were done in this group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- crestal technique using densah burs (Experimental): Seven implant sites underwent sinus membrane elevation procedure using densah burs with crestal approach. Crestal flap was made and Densah bur with diameter 2.00 mm will be used in osseodensification mode with copious irrigation till sinus floor, then diameter 3.00 mm bur up to 3 mm past the sinus floor, then sequential wider burs to reach the final desired width followed by bone grafting and simultaneous implant placement.
  Interventions: Procedure: crestal sinus lifting using densah burs
- lateral window technique (Active Comparator): Seven implant sites underwent sinus membrane elevation procedure using lateral window technique. Pyramidal flap was made and an trap door is created in the lateral sinus wall to gain access to Schneiderian membrane in order to elevate it and provide space for the bone graft material to be placed followed by simultaneous implant placement.
  Interventions: Procedure: sinus lifting using lateral window technique

INTERVENTIONS:
Procedure: crestal sinus lifting using densah burs — * Crestal flap was made.
  * 2 mm densah bur was used first as a pilot drill in clockwise direction and stopped 1 mm before sinus floor. Implant surgical motor setting was changed to reverse.
  * The next wider densah bur (3.00 mm) was used and advanced into the previous created osteotomy. When feeling the haptic feedback of the bur reaching the dense sinus floor, pressure was modulated with a pumping motion to advance past the sinus floor in 1 mm increments, up to 3 mm.
  * The sequential wider densah burs were used in densifing mode with copious irrigation with pumping motion to achieve additional width with maximum membrane lift of 3 mm to reach final desired width for implant placement.
  * The osteotomy was filled with a well hydrated, xenograft. The last densah bur was used in densifing mode with low speed 150-200 rpm with no irrigation.
  * The implant was placed into the osteotomy.
  Arms: crestal technique using densah burs
Procedure: sinus lifting using lateral window technique — * Trapezoidal flap was made and full thickness mucoperiosteal flap was raised to visualize the lateral side of the maxilla. (Fig. 23)
  * Complete osteotomy of lateral window was made to gain access to the Schneiderian membrane using piezosurgery unit to minimize the probability of membrane perforation with round tip (SL3).
  * Sinus membrane elevators were used carefully to free up sinus membrane in all directions (mesially, distally and medially).
  * The membrane at the inferior aspect of the osteotomy was dissected from the floor of the maxillary sinus and elevated upward to create a space in the floor of the sinus for the bone graft material.
  * Drilling of the implant was done using surgical implant kit while using periosteal elevators to protect schniderian membrane.
  * Bone graft was packed under the membrane in all directions with the help of pluggers till reach the medial wall of the maxillary sinus.
  * Implant was placed and the lateral osteotomy was covered with collagen membrane
  Other Names: lateral sinus lifting
  Arms: lateral window technique

SUMMARY:
The aim of the study was to assess the clinical and radiographic outcomes of crestal sinus lifting using densah burs versus lateral window technique in vertically deficient posterior maxilla with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient medically free from systemic, immunologic or debilitating diseases or local conditions that could affect normal bone healing and/or implant placement.

  2. Patient with good oral hygiene. 3. Age from 18 to 55 years. 4. Partially edentulous patients with missed one or more of maxillary posterior teeth with residual alveolar ridge height 3-5 mm and a minimal width of the alveolar ridge 7 mm in the region of the planned implant site.

  5. Patients' edentulous ridges covered with optimal width of keratinized mucosa (<3 mm) with no signs of inflammation, ulceration of scar tissue.

  6. No history of parafunctional habits. 7. Patients were ready to comply with the follow-up and maintenance program. 8. Sufficient inter arch space for prothesis.

Exclusion Criteria:

- 1. Patients with clinical or radiographic evidence of rhinosinusitis or any other pathology in the maxillary sinus.

2. Smokers. 3. Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
change from baseline in pain, as measured by Numerical Rating Scale (NRS) | Baseline, 7 days
  Pain was evaluated postoperatively at the day of surgery, 3rd and 7th day post-surgically Numerical Rating Scale (NRS). Numerical Rating Scale (NRS) is a simple, widely used tool, typically an 11-point scale (0-10), where patients rate their pain intensity, with 0 meaning "no pain" and 10 meaning "worst imaginable pain,".
change from baseline of edema | baseline, 7 days
  Edema was evaluated with the aid of tape measure (in centimeters). Three measurements were performed on the patient's operated site preoperatively, 3rd and 7th day after surgery. The evaluation of edema was done by subtracting the total value of the three measurements obtained postoperatively (at 3rd and 7th day) from the total value of the three measurements obtained at pre-operative baseline.
  The three measuring lines are:
  1. Lateral corner of the eye-angle of the mandible.
  2. Tragus-outer corner of the mouth.
  3. Tragus pogonion.
change of implant stability, as measured by osstell | baseline, 12 months
  Stability was measured with osstell (ISQ) immediately after implant placement (T0) after 12 months (T12). ISQ is a scale that ranges from 1 to 100 and is used to assess implant stability. Scales greater than 70 ISQ indicate a high level of stability, scales between 60 and 69 means medium stability and scales >60 ISQ are considered as low stability.
change from baseline in Grafted sinus height (GSH) | baseline, 12 months
  CBCT was made preoperatively, immediately after sinus augmentation (T0) and 6 months after loading (T12) for evaluation of Grafted sinus height (GSH): the distance between the original sinus floor to the new sinus floor regarding crestal cortical line.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Mohamed Ahmed, professor, Study Director — department of oral and maxillofacial surgery, faculty of dentistry, mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No